CLINICAL TRIAL: NCT02375828
Title: Tolerance and Acceptability of Glibentek in Patients With Neonatale Diabetes Secondary to Mutations in K+-ATP Channels
Brief Title: Glibentek in Patients With Neonatal Diabetes Secondary to Mutations in K+-ATP Channels
Acronym: NEOGLI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-003436-39
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neonatal Diabetes Secondary to Mutation in the Potassium Channel
Keywords: Acceptability; Phase 3; Neonatal diabetes
MeSH Terms: interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with neonatal diabetes (Experimental): Patients with neonatal diabetes
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Glibenclamide — Glibenclamide pills will be administrated during one month at the previously used dosage. During the first month of the study we wwil record pharmacokinetic data, number of hypoglycaemia and the administration problems associated to this galenic form. At the end of the first month of enrolment, patients will be given oral solution of glibenclamide for the 4 remaining months. Pharmacocinetic data, number of hypoglycaemia and parents and children feeling about pratictability of administration will be then recorded.

SUMMARY:
The understanding of the molecular mechanisms of neonatal diabetes has deeply changed the therapy of patients carrying mutations in the K-ATP channel. Indeed, those patients are not treated anymore by insulin injections but by glibenclamide an oral anti-diabetic drug widely used in type 2 diabetes. Anyway, its galenic form (pills of 5 mg) is not suitable for children and difficult to administrate to infants or young children. The purpose of this study is to determine if a new galenic form of this durg is more suitable and as efficient as pills in children with neonatal diabetes.

DETAILED DESCRIPTION:
Neonatal diabetes mellitus (NDM), characterized by hyperglycaemia requiring exogenous insulin therapy, is a rare condition that appears during the first months of life with an estimated incidence of 1 in 12000 newborns. We recently published that in our large cohort, the origin of the disease is an heterozygous activating mutation of the coding sequence of KCNJ11 or ABCC8 genes in 42% of patients. These genes encode for the Kir 6.2 subunit (KCNJ11 gene) and for the SUR1 subunit (ABCC8 gene) of the ATP-sensitive K+ channel (KATP) whom function in the beta cell is to induce a membrane depolarization triggering the exocytosis of insulin-containing granules. The understanding of the molecular substrate of the disease has deeply changed the therapy, allowing the switch from insulin injections to an oral medication with sulfonylureas. Indeed, these drugs specifically bind to SUR1 subunit increasing the closing ability of the KATP by an ATP-independent mechanisms stimulating insulin secretion. Together with others we demonstrated that these drugs were efficient in replacement of subcutaneous injected insulin in children or adults with a Kir6.2 or a SUR1 activating mutation allowing an excellent metabolic control of the disease without the side effects of insulin (hypoglycemia).

Anyway, in most countries, glibenclamide has not been approved for use in children by heath authorities in france and its use is then only temporary tolerated in this specific indication.

Furthermore its galenic form (pills) is not suitable for children and especially for infants. The dosage is too high for most infants and young children or children wih neurologic defects (frequently associated to this kind of neonatal diabetes) can't swallow pills. Chewing the pill can't be an alternative as sulfamides are known induce alterations of tooth enamel color.

Most patients parents have to crush the pills and dilute the powder in water before administrating it to their child. Such process doesn't follow recommendations of administration of and medicine contradiction. It can also alter the drug cinetic.as glibenclamide is not completely soluble in water.

After our successful clinical trial, we decided then to be a part in the development of a galenice form suitable for children. The AMMtek company has created a new galenic dedicated to pediatric patients. This new oral solution has been demonstrated to be safe and effective in a phase 1 study. Its pediatric investigation plan has been validated in july 2013 by the European medicine agency. The French drug and food agency (ANSM) has asked for a tolerance and acceptability study before giving its approval for use in children and infants with neonatal diabetes.

The aim of this study is then to determine the tolerance and acceptability of an oral solution of glibenclamide (Glinbentek) developed and dedicated to pediatric patients with neonatal diabetes secondary to mutation in potassium channels.

ELIGIBILITY:
Inclusion Criteria:

* Age below 18 years
* Neonatal diabetes secondary to documented mutation in one of the 2 sub units of potassium channels
* Patients already treated by glibenclamide pills
* Signed consent

Exclusion Criteria:

* Families unable to fill in the questionnaries
* Patients unable to answer to the visual hedonic squale
* Patients unable to take the oral solution
* Known allergy to sulfonylureas or to other antidiabetic or antibiotic sulfamides
* Insulin therapy associated to glibenclamide
* Miconazole therapy
* Porphyria
* Breast feeding
* Severe renal failure (creatinine clearance below 30 ml/mn)
* Liver failure (prothombine time below 70)
* Not affiliated to the health care system

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Acceptability of an oral solution of glibenclamide (Hedonic visual scale) | 2 months after the change from pills to oral solution.
  Hedonic visual scale
Acceptability of an oral solution of glibenclamide (Hedonic visual scale) | 3 months after the change from pills to oral solution.
  Hedonic visual scale

SECONDARY OUTCOMES:
Tolerance of an oral solution of glibenclamide (Self administrated questionnaries) | 2 months after the change from pills to oral solution.
  Self administrated questionnaries, liver and renal biology
Tolerance of an oral solution of glibenclamide (Self administrated questionnaries) | 3 months after the change from pills to oral solution.
  Self administrated questionnaries, liver and renal biology
Recording pharmaceutical data on pills and oral solution of glibenclamide (Blood drug dosage) | At inclusion
  Blood drug dosage
Recording pharmaceutical data on pills and oral solution of glibenclamide (Blood drug dosage) | 2 months after the switch from pills to oral solution
  Blood drug dosage
No alteration in metabolic control of the disease | During the first month of administration
  HbA1C at month 3, fructosamine at month 2 and 3, self record of hypoglycaemia during month 1, 2 and 3, glycemia before and after meals during 2 consecutive days at introduction of oral solution and during 2 meals at month 2 and month 3
No alteration in metabolic control of the disease | 2 months after the change from pills to oral solution
  HbA1C at month 3, fructosamine at month 2 and 3, self record of hypoglycaemia during month 1, 2 and 3, glycemia before and after meals during 2 consecutive days at introduction of oral solution and during 2 meals at month 2 and month 3
No alteration in metabolic control of the disease | 3 months after the change from pills to oral solution
  HbA1C at month 3, fructosamine at month 2 and 3, self record of hypoglycaemia during month 1, 2 and 3, glycemia before and after meals during 2 consecutive days at introduction of oral solution and during 2 meals at month 2 and month 3

CONTACTS AND LOCATIONS:
Overall Officials: Michel Polak, MD, PhD, Study Director — Hopital Universitaire Necker Enfants Malades, Assistance publique - hôpitaux de Paris, Faculté de medicine Paris Descartes, Université Sorbonne Paris cité
Locations (1):
- Hôpital Universitaire Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Beltrand J, Baptiste A, Busiah K, Bouazza N, Godot C, Boucheron A, Djerada Z, Gozalo C, Berdugo M, Treluyer JM, Elie C, Polak M; GLID-KIR study group. Glibenclamide oral suspension: Suitable and effective in patients with neonatal diabetes. Pediatr Diabetes. 2019 May;20(3):246-254. doi: 10.1111/pedi.12823. Epub 2019 Feb 21. PMID 30684309
- [Background] Busiah K, Drunat S, Vaivre-Douret L, Bonnefond A, Simon A, Flechtner I, Gerard B, Pouvreau N, Elie C, Nimri R, De Vries L, Tubiana-Rufi N, Metz C, Bertrand AM, Nivot-Adamiak S, de Kerdanet M, Stuckens C, Jennane F, Souchon PF, Le Tallec C, Desiree C, Pereira S, Dechaume A, Robert JJ, Phillip M, Scharfmann R, Czernichow P, Froguel P, Vaxillaire M, Polak M, Cave H; French NDM study group. Neuropsychological dysfunction and developmental defects associated with genetic changes in infants with neonatal diabetes mellitus: a prospective cohort study [corrected]. Lancet Diabetes Endocrinol. 2013 Nov;1(3):199-207. doi: 10.1016/S2213-8587(13)70059-7. Epub 2013 Sep 6. PMID 24622368
- [Background] Pearson ER, Flechtner I, Njolstad PR, Malecki MT, Flanagan SE, Larkin B, Ashcroft FM, Klimes I, Codner E, Iotova V, Slingerland AS, Shield J, Robert JJ, Holst JJ, Clark PM, Ellard S, Sovik O, Polak M, Hattersley AT; Neonatal Diabetes International Collaborative Group. Switching from insulin to oral sulfonylureas in patients with diabetes due to Kir6.2 mutations. N Engl J Med. 2006 Aug 3;355(5):467-77. doi: 10.1056/NEJMoa061759. PMID 16885550
- [Background] Babenko AP, Polak M, Cave H, Busiah K, Czernichow P, Scharfmann R, Bryan J, Aguilar-Bryan L, Vaxillaire M, Froguel P. Activating mutations in the ABCC8 gene in neonatal diabetes mellitus. N Engl J Med. 2006 Aug 3;355(5):456-66. doi: 10.1056/NEJMoa055068. PMID 16885549